CLINICAL TRIAL: NCT05397132
Title: Mechanisms of Disease Relapse/Resistance in CAR T Therapy for Hematologic Malignancies
Brief Title: Mechanisms of Disease R/R in CAR-T for Hematologic Malignancies
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00109903; 1R21CA267275-01 (NIH)
Record Dates: First submitted 2022-05-11; First posted 2022-05-31 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Malignancy
Keywords: CAR-T
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood for banking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Blood draw — Patients will provide a blood draw for research and repository

SUMMARY:
The primary purpose of this IRB protocol is to perform immune profiling focusing on the measurement of Myeloid derived suppressor cells (MDSCs) over time in patients receiving Chimeric antigen receptor (CAR) T therapy and determine the correlation between immune profile and disease relapse/resistance in CAR T therapy.

DETAILED DESCRIPTION:
The primary purpose of this IRB protocol is to perform immune profiling focusing on the measurement of MDSCs over time in patients receiving CAR T therapy and determine the correlation between immune profile and disease relapse/resistance in CAR T therapy. Blood samples and accompanying health information (including PHI) may be collected from standard of care, non-significant risk, research-only procedures or obtained from our Division Research Repository and Database (Duke IRB Pro00006268) or DUHS Biospecimen Research and Biobanking protocol (Duke IRB Pro00035974). All hematologic malignancy patients treated with commercial CAR T products will be screened and enrolled for the study.

The investigators will perform multivariable regression to see if the number and function of MDSCs can be used as independent factors to predict disease relapse at 1 year after CAR T treatment, overall survival or progression-free survival. The studies will not require additional invasive procedure solely for the study.

The investigators will use blood samples that are performed as part of standard care. Therefore, no additional procedure is needed. The major potential risk associated with the study is the breach of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and provide signed informed consent that fulfills Institutional Review Board guidelines.
2. Has a confirmed diagnosis of hematologic malignancy and will be undergoing CAR T therapy with commercial CAR T product.
3. Patient who has a confirmed diagnosis of hematologic malignancy and will be receiving CAR T therapy under clinical trial protocol will also be eligible if the clinical trial sponsor and the investigator approve patient participation in the study.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between change in immune profile and disease relapse/resistance in CAR T therapy | before CAR T therapy, 1 week after CAR T and then every 3-6 months, and at the time of disease relapse (up to 5 years)
  multivariable regression

SECONDARY OUTCOMES:
Correlation between change in molecular/genetic analysis and disease relapse/resistance in CAR T therapy | before CAR T therapy, 1 week after CAR T and then every 3-6 months, and at the time of disease relapse (up to 5 years)
  bulk RNA-sequencing, single cell RNA sequencing, single cell ATAC seq or metabolomics on peripheral blood samples
Correlation between changes in cytokine and molecular pathway profiling with disease relapse/resistance in CAR T therapy | before CAR T therapy, 1 week after CAR T and then every 3-6 months, and at the time of disease relapse (up to 5 years)
  Cytokine profiling and molecular/genetic correlation with disease relapse/resistance in CAR T therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yubin Kang, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No